CLINICAL TRIAL: NCT01266694
Title: Cochicine Treatment for Post- Operative Pericardial Effusion: The POPE 2 Study A Multicenter, Double-blind, Randomized Trial
Brief Title: Cochicine Treatment for Post- Operative Pericardial Effusion
Acronym: POPE2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: French Federation of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-02
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Pericardial Effusion
Keywords: Pericardial effusion; Cardiac surgery; Tamponade; colchicine
MeSH Terms: conditions — Pericardial Effusion | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cochicine (Experimental): Colchicine arm: patient receiving 1 mg per day for 14 days
  Interventions: Drug: Colchicines
- Placebo (Placebo Comparator): patients placebo controlled
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicines — oral form, 1 mg, once a day during 14 days
  Arms: Cochicine
Drug: Placebo — oral form, placebo
  Arms: Placebo

SUMMARY:
Background: The incidence of asymptomatic pericardial effusion is high after cardiac surgery.

Objective: To assess whether colchicine is effective in reducing post operative pericardial effusion volume.

Design: Multicenter, randomized, double-blind, placebo-controlled study. Intervention : colchicine 1mg vs placebo, once daily for 14 days Setting :10 post operative cardiac rehabilitation centers. Patients: 200 patients at high risk of tamponade because of moderate to large persistent pericardial effusion (grade 2, 3 or 4 on a scale of 0 to 4 measured by echocardiography) more than 7 days after cardiac surgery.

Measurements: The main end point will be change in effusion grade after 14 days of treatment. Secondary endpoints include frequency of late cardiac tamponade.

DETAILED DESCRIPTION:
Clinically insignificant pericardial effusion is common after heart surgery with an incidence of 50 % to 85 % a few days after surgery Cardiac tamponade occurs in about 1-2 % of patients who undergo cardiac surgery and may develop slowly without clear-cut clinical signs. Most tamponade occurs more than 7 days after surgery which is a concern because, at that time, patients often have already been discharged from the hospital.

No study has ever shown the efficacy any drug for this condition.In particular, we published a study demonstrating the absence of efficacy of a non steroidal anti inflammatory drug (Meurin P, Tabet JY, Thabut G, et al.French Society of Cardiology. Nonsteroidal anti-inflammatory drug treatment for postoperative pericardial effusion: a multicenter randomized, double-blind trial. Ann Intern Med. 2010 Feb2;152(3):137-43) Cochicine is widely used to treat inflammatory pericarditis ; is it efficient to treat post operative pericardial effusions ? this is the question we want to answer to.

Design: Multicenter, randomized, double-blind, placebo-controlled study. Intervention : colchicine 1mg vs placebo, once daily for 14 days Setting :10 post operative cardiac rehabilitation centers. Patients: 200 patients at high risk of tamponade because of moderate to large persistent pericardial effusion (grade 2, 3 or 4 on a scale of 0 to 4 measured by echocardiography) more than 7 days after cardiac surgery.

Measurements: The main end point will be change in effusion grade after 14 days of treatment. Secondary endpoints include frequency of late cardiac tamponade.

ELIGIBILITY:
Inclusion Criteria:

* patients with recent cardiac surgery
* admitted for cardiac rehabilitation
* pericardial effusion > grade 2 (corresponds to a loculated effusion > 10 millimeters or a circumferential effusion of any size)on the first trans thoracic echocardiography performed more than 7 days after surgery

Exclusion Criteria:

* patients who do not give written consent to participate
* pregnancy
* colchicine allergy;
* renal failure, which we define as a serum creatinine level > 250micromol/l or clairance < 30 ml/mn
* heart transplantation,or correction of congenital heart anomalies cardiac surgery more than 30 days before their first trans thoracic echocardiography pericardial effusion that requires immediate drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
change in effusion grade | 14 days

SECONDARY OUTCOMES:
frequency of late cardiac tamponade | 14 days
number of patients with at least a one-grade decrease in the effusion | 14 days
mean change in the width of the effusion measured in millimeters | 14 days
evolution of prespecified subgroups | 14 days
  * patients with inflammatory syndrom : crp > 30 mg/l
  * patients receiving an anticoagulant
  * patients with a post pericardiotomy syndrom

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Meurin, MD, Principal Investigator — Clinique Les Grands Près - Villeneuve Saint Denis
Locations (10):
- France (10):
  - Bois Gibert, Ballan-Miré
  - Centre Médical de Bligny, Briis-sous-Forges
  - Clinique de Châtillon, Châtillon
  - Centre Dieulefit Santé, Dieulefit
  - Hopital Corentin Celton, Issy-les-Moulineaux
  - Clinique de la mitterie, Lomme
  - Centre Hospitalier Loire Vendée Océan, Machecoul
  - Clinique Iris, Marcy-l'Étoile
  - Maison du mineur, Vence
  - Clinique les Grands Près, Villeneuve-Saint-Denis

REFERENCES:
- [Derived] Meurin P, Lelay-Kubas S, Pierre B, Pereira H, Pavy B, Iliou MC, Bussiere JL, Weber H, Beugin JP, Farrokhi T, Bellemain-Appaix A, Briota L, Tabet JY; French Society of Cardiology. Colchicine for postoperative pericardial effusion: a multicentre, double-blind, randomised controlled trial. Heart. 2015 Nov;101(21):1711-6. doi: 10.1136/heartjnl-2015-307827. Epub 2015 Jun 15. PMID 26076938